CLINICAL TRIAL: NCT01558258
Title: A Mindfulness Meditation-Based Intervention for Younger Breast Cancer Survivors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 10-001799; SAC110009 (Other: Susan G. Komen Foundation)
Record Dates: First submitted 2012-02-17; First posted 2012-03-20 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Younger Breast Cancer Survivors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfullness Meditation-based Intervention (Experimental): Mindfulness meditation-based intervention, is a 6-week program adapted from an existing program at Mindfulness Awareness Research Center(MARC),UCLA.
  Interventions: Behavioral: Mindful Awareness practices (MAPs)
- Wait-list control group (No Intervention): The wait-list control condition will control for naturally occurring changes in stress and other outcomes over the six-week intervention period. After the post-treatment assessments have been completed, those assigned to the wait-list control group will be able to participate in the MAP classes.

INTERVENTIONS:
Behavioral: Mindful Awareness practices (MAPs) — Mindfulness meditation-based intervention, is a 6-week program adapted from an existing program at Mindfulness Awareness Research Center(MARC),UCLA.
  Arms: Mindfullness Meditation-based Intervention

SUMMARY:
Younger women with breast cancer experience substantially greater distress and depressive symptoms than older women. These symptoms can hamper recovery and healthy behaviors that can reduce the risk of recurrence and/or other chronic diseases. The primary objective of this study is to evaluate the feasibility and preliminary efficacy of a mindfulness meditation-based intervention for this at-risk group of women. The investigators hypothesize that a structured program of mindfulness meditation will lead to significant improvements in psychological well-being (i.e., depression, stress), with corresponding improvements in health behaviors and biomarkers of cancer risk, in women diagnosed with breast cancer, prior to age 50. The investigators will also examine mechanisms for intervention effects, including increased mindfulness and ability to relax.

ELIGIBILITY:
Inclusion Criteria:

* women diagnosed with early, resectable breast cancer (Stage 0, I, II, or III) prior to age 50
* have completed treatment with surgery, radiation, and/or chemotherapy at least 3 months previously.

Exclusion Criteria:

* have a breast cancer recurrence, metastasis, or another cancer diagnosis (excluding non-melanoma skin cancer
* unable to commit to intervention schedule.

Max Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 71 (Actual)
Dates: Start 2011-04; Primary Completion 2014-02 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Effect of Mindful Awareness Practices on daily living. | 6 weeks
  Participants meet for 6 weekly, 2hr group sessions that include presentation of theoretical materials on mindfulness,relaxation,and mind-body connection;experiential practice of meditation and gentle yoga;psycho-educational component for cancer survivors,and group process focused on solving problems concerning impediments to effective practice.Participants will be instructed to practice mindfulness techniques on a daily basis. Daily diaries will be kept by participants to record practice time, mood assessments, and self-reported questions on benefits and barriers to practicing.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Ganz, M.D., Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA, Los Angeles, California, United States